CLINICAL TRIAL: NCT00000311
Title: Combining Behavioral Treatment With Agonist Maintenance
Brief Title: Combining Behavioral Treatment With Agonist Maintenance - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Richard S. Schottenfeld, MD, Yale University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09413-1; R01DA009413 (NIH); R01-09413-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Cocaine-Related Disorders; Opioid-Related Disorders; Substance-Related Disorders
Keywords: Cocaine-Related Disorders; Opioid-Related Disorders; Substance-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine; Methadone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 (Experimental): Methadone + CM (contingency management)
  Interventions: Drug: methadone
- 2 (Experimental): methadone + VC (voucher control)
  Interventions: Drug: methadone
- 3 (Experimental): Buprenorphine + CM
  Interventions: Drug: Buprenorphine
- 4 (Experimental): Buprenorphine + VC
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Medication and Behavioral
  Arms: 3; 4
Drug: methadone — medication and behavioral
  Arms: 1; 2

SUMMARY:
The purpose of this study is to evaluate whether the community reinforcement approach (CRA) plus contingency management (CM) is more effective overall than CRA only in reducing illicit opioid and cocaine use during agonist maintenance treatment and at 3 and 6 month follow-up after completion of study protocol, and to compare the efficacy of maintenance on buprenorphine to methadone when maintenance is combined with CRA only or CRA plus CM.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 1995-02; Primary Completion 1999-02 (Actual); Study Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
Depression | 24 weeks
Withdrawal symptoms
Opioid and cocaine use
Social and psychological functioning
AIDS risk behavior

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schottenfeld, M.D., Principal Investigator — Yale University
Locations (1):
- APT Residential Services Division, New Haven, Connecticut, United States